CLINICAL TRIAL: NCT00933985
Title: A Phase I Study of Obatoclax (Pan Anti-Apoptotic BCL-2 Family Small Molecule Inhibitor), in Combination With Vincristine/Doxorubicin/Dexrazoxane, in Children With Relapsed/Refractory Solid Tumors or Leukemia
Brief Title: Obatoclax Mesylate, Vincristine Sulfate, Doxorubicin Hydrochloride, and Dexrazoxane Hydrochloride in Treating Young Patients With Relapsed or Refractory Solid Tumors, Lymphoma, or Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01936; NCI-2011-01936 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL0816; CDR0000647160; ADVL0816 (Other: COG Phase I Consortium); ADVL0816 (Other: CTEP); U01CA097452 (NIH)
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Acute Leukemias of Ambiguous Lineage; Acute Undifferentiated Leukemia; Angioimmunoblastic T-cell Lymphoma; Blastic Phase Chronic Myelogenous Leukemia; Childhood Burkitt Lymphoma; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Relapsing Chronic Myelogenous Leukemia; Small Intestine Lymphoma; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Immunoblastic Lymphadenopathy; Blast Crisis; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Extranodal NK-T-Cell; Intraocular Lymphoma; Lymphoma, T-Cell, Peripheral; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell | interventions — Dexrazoxane; Razoxane; Doxorubicin; obatoclax; Vincristine

ARMS (1):
- Treatment (obatoclax, vincristine, doxorubicin, dexrazoxane) (Experimental): STRATUM 1 (dose-escalation): Patients receive obatoclax mesylate IV over 3 hours on days 1 and 8 and vincristine sulfate IV, doxorubicin hydrochloride IV, and dexrazoxane hydrochloride IV on day 8 of course 1 (28 days). Drugs are administered on day 1 of subsequent courses and repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  STRATUM 2: Patients receive obatoclax mesylate (at starting dose in stratum 1), vincristine sulfate, doxorubicin hydrochloride, and dexrazoxane hydrochloride as in stratum 1.
  STRATUM 3: Patients receive obatoclax mesylate (at the MTD determined in stratum 1), vincristine sulfate, doxorubicin hydrochloride, and dexrazoxane hydrochloride as in stratum 1.
  Interventions: Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: obatoclax mesylate; Drug: liposomal vincristine sulfate; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: dexrazoxane hydrochloride — Given IV
  Other Names: Cardioxane; Savene; Totect; Zinecard
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: obatoclax mesylate — Given IV
  Other Names: GX15-070MS
Drug: liposomal vincristine sulfate — Given IV
  Other Names: liposomal vincristine; Marqibo; vincristine liposomal; vincristine sulfate liposome injection
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of obatoclax mesylate when given together with vincristine sulfate, doxorubicin hydrochloride, and dexrazoxane hydrochloride in treating young patients with relapsed or refractory solid tumors, lymphoma, or leukemia. Obatoclax mesylate may stop the growth of cancer cells by blocking some of the proteins needed for cell growth and causing the cells to self-destruct. Drugs used in chemotherapy, such as vincristine sulfate, doxorubicin hydrochloride, and dexrazoxane hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving obatoclax mesylate together with combination chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended Phase II dose of obatoclax (obatoclax mesylate) administered as a single agent on day 1 and in combination with vincristine ( vincristine sulfate), doxorubicin (doxorubicin hydrochloride), and dexrazoxane (dexrazoxane hydrochloride) at day 8 in children with refractory solid tumors.

II. To define and describe the toxicities of obatoclax administered on this schedule.

III. To characterize the pharmacokinetics of obatoclax in children with refractory solid tumors or relapsed leukemia.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of obatoclax in children with refractory or relapsed solid tumors and leukemias within the confines of a Phase I study.

II. To preliminarily assess leukemic blast characteristics associated with obatoclax activity.

III. To preliminarily assess the biological activity of obatoclax by investigating effects on cell death regulatory pathways.

OUTLINE: This is a dose-escalation study of obatoclax mesylate.

STRATUM 1 (dose-escalation): Patients receive obatoclax mesylate intravenously (IV) over 3 hours on days 1 and 8 and vincristine sulfate IV, doxorubicin hydrochloride IV, and dexrazoxane hydrochloride IV on day 8 of course 1 (28 days). Drugs are administered on day 1 of subsequent courses and repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

STRATUM 2: Patients receive obatoclax mesylate (at starting dose in stratum 1), vincristine sulfate, doxorubicin hydrochloride, and dexrazoxane hydrochloride as in stratum 1.

STRATUM 3: Patients receive obatoclax mesylate (at the MTD determined in stratum 1), vincristine sulfate, doxorubicin hydrochloride, and dexrazoxane hydrochloride as in stratum 1.

After completion of study therapy, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Stratum 1 (solid tumors, including lymphomas): patients must have had histologic verification of malignancy at original diagnosis or relapse; patients with recurrent or refractory solid tumors are eligible, excluding primary central nervous system (CNS) tumors or patients with known CNS metastases
* Stratum 2 (mixed-lineage leukemia [MLL] + leukemia): patients with recurrent or refractory MLL+ leukemia are eligible excluding those patients with symptomatic CNS leukemia, CNS chloromas, or leptomeningeal leukemic involvement
* Stratum 3 (other leukemias): patients with non-MLL+ recurrent or refractory leukemia (acute lymphoblastic leukemia [ALL], acute myeloid leukemia [AML] or chronic myeloid leukemia [CML] in blast crisis) are eligible excluding those patients with symptomatic CNS leukemia, CNS chloromas, or leptomeningeal leukemic involvement
* Stratum 1: patients must have either measurable or evaluable disease
* Strata 2 and 3: patients with leukemia must have a > 25% blasts on bone marrow aspirate to be eligible
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  * Myelosuppressive chemotherapy: must not have received within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea); hydroxyurea may be administered prior to study enrollment; in such cases at least 24 hours must have elapsed between the last dose of hydroxyurea and the first dose of obatoclax
  * Hematopoietic growth factors: at least 7 days since the completion of therapy with a growth factor
  * Biologic (anti-neoplastic agent): at least 7 days since the completion of therapy with a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * Immunotherapy: at least 6 weeks since the completion of any type of immunotherapy, e.g. tumor vaccines
  * Monoclonal antibodies: at least 3 half-lives since prior therapy that includes a monoclonal antibody
  * Radiation therapy (XRT): >= 2 weeks (wks) for local palliative XRT (small port); >= 6 months must have elapsed if prior total-body irradiation (TBI), craniospinal XRT or if >= 50% radiation of pelvis; >= 6 wks must have elapsed if other substantial bone marrow (BM) radiation
  * Stem cell transplant or rescue without TBI: no evidence of active graft vs. host disease and >= 3 months must have elapsed since transplant
* STRATUM 1: Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* STRATUS 1: Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
* STRATUM 1: Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* STRATA 2 and 3: Platelet count >= 20,000/mm^3 (may receive platelet transfusions)
* STRATA 2 and 3: Hemoglobin >= 8.0 g/dL (may receive RBC transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70ml/min/1.73 m^2 OR a serum creatinine based on age/gender as follows:

  * 0.5 mg/dL (6 months to < 1 year of age)
  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (>= 16 years of age)
* Bilirubin (sum of conjugated + unconjugated) >= 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) >= 110 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin >= 2 g/dL
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by gated radionuclide study
* Stable neurological examination for at least 2 weeks prior to study enrollment; no known > grade 2 unresolved neurological toxicities
* All patients and/or their parents or legal guardians must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Growth factors that support platelet or white cell number or function must not have been administered within the 7 days prior to enrollment
* Patients requiring corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the prior 7 days
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anticancer agents, with the exception of hydroxyurea, are not eligible; patients with leukemia may receive intrathecal therapy as outlined
* Any anti-convulsant medications
* Patients who have an uncontrolled infection are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* Patients with a total lifetime cumulative anthracycline dose > 750 mg/m2 (25 mg/kg if < 1 year) doxorubicin or equivalent at the time of enrollment are not eligible

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2009-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose of obatoclax mesylate in combination with vincristine sulfate, doxorubicin hydrochloride, and dexrazoxane hydrochloride, defined as the maximum dose at which fewer than one-third of patients experience dose limiting toxicity | 28 days
  Will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0).
Incidence of adverse events characterized by grade, relationship to study therapy, and prior experience, assessed by NCI CTCAE v4.0 | Up to 30 days
  Descriptive summary of all toxicities will be reported.

SECONDARY OUTCOMES:
Disease response assessed using Response Evaluation Criteria in Solid Tumors | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aplenc, Principal Investigator — COG Phase I Consortium
Locations (20):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Childrens Hospital of Orange County, Orange, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Derived] Urtishak KA, Edwards AY, Wang LS, Hudome A, Robinson BW, Barrett JS, Cao K, Cory L, Moore JS, Bantly AD, Yu QC, Chen IM, Atlas SR, Willman CL, Kundu M, Carroll AJ, Heerema NA, Devidas M, Hilden JM, Dreyer ZE, Hunger SP, Reaman GH, Felix CA. Potent obatoclax cytotoxicity and activation of triple death mode killing across infant acute lymphoblastic leukemia. Blood. 2013 Apr 4;121(14):2689-703. doi: 10.1182/blood-2012-04-425033. Epub 2013 Feb 7. PMID 23393050